CLINICAL TRIAL: NCT02350686
Title: Phase II Study of Second Line Capecitabine Plus Oxaliplatin (XELOX) in Patients With Advanced Biliary Tract Carcinoma After Failure of Gemcitabine-based Chemotherapy
Brief Title: XELOX in Advanced Biliary Tract Carcinoma After Failure of Gemcitabine-based Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, MD, PhD, Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-09-020
Record Dates: First submitted 2014-11-24; First posted 2015-01-30 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capecitabine+oxaliplatin (Experimental): XELOX every 3 weeks
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — XELOX every 3 weeks will be continued until disease progression, patients' refusal or upto 8 cycles
  Other Names: xeloda
Drug: oxaliplatin — XELOX every 3 weeks will be continued until disease progression, patients' refusal or upto 8 cycles

SUMMARY:
Phase II study of second line capecitabine plus oxaliplatin (XELOX) in patients with advanced biliary tract carcinoma after failure of gemcitabine-based chemotherapy.

DETAILED DESCRIPTION:
XELOX

* Xeloda, 1000mg/㎡ bid, day 1-15, every 3 weeks
* Oxaliplatin 130mg/㎡, day 1, every 3 weeks Until disease progression, patient's refusal or up to 8 cycles (maximum).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. histologically or cytologically confirmed adenocarcinoma of biliary tract (intrahepatic, extrahepatic cholangiocarcinoma, gall bladder cancer and ampulla of Vater cancer)
3. unresectable or metastatic
4. progression after treatment with first line gemcitabine-based chemotherapy
5. ECOG performance status of 0~2
6. measurable or evaluable lesion per RECIST 1.1 criteria
7. adequate marrow, hepatic, renal and cardiac functions

Exclusion Criteria:

1. severe co-morbid illness or active infections
2. pregnant or lactating women
3. History of documented congestive heart failure, angina pectoris requiring medication, evidence of tranasmural myocardial infarction on ECG, poorly controlled hypertension, clinically significant valvular heart disease or high risk of uncontrollable arrhythmia
4. active CNS metastases not controllable with radiotherapy or corticosteroids
5. known history of hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2015-05-14 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12months

SECONDARY OUTCOMES:
response rate | 12months
duration of response | 12months
overall survival | 12months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea